CLINICAL TRIAL: NCT06254898
Title: Use of Incentives for Children Undergoing Stressful Medical Procedures
Brief Title: Use of Incentives for Stressful Medical Procedures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jennifer Staab, MS, CCLS (Other)
Responsible Party: Sponsor-Investigator, Jennifer Staab, MS, CCLS, Principal Investigator, Children's Hospital Colorado
Organization: Children's Hospital Colorado (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 23-0337
Record Dates: First submitted 2023-12-07; First posted 2024-02-12 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: pediatrics; child life; medical procedures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Child life standard of care (Active Comparator): Child life standard of care
  Interventions: Behavioral: Child life standard of care
- Child life standard of care + incentives provided with conditional agreement. (Experimental): Child life standard of care + incentives provided with conditional agreement.
  Interventions: Behavioral: Child life standard of care + incentives provided with conditional agreement.
- Child life standard of care + incentive provided unconditionally. (Experimental): Child life standard of care + incentive provided unconditionally.
  Interventions: Behavioral: Child life standard of care + incentive provided unconditionally.

INTERVENTIONS:
Behavioral: Child life standard of care — Standard preparation and support provided to the participant by a Certified Child Life Specialist.
  Arms: Child life standard of care
Behavioral: Child life standard of care + incentives provided with conditional agreement. — Patient is provided standard preparation and support provided to the participant by a Certified Child Life Specialist. Before the procedure the child life specialist discusses earning a prize with the patient if they demonstrate the agreed upon coping goal (i.e. holding arm still, taking deep breaths, engaging in distraction.) At the end of the procedure the patient is provided with the prize if they earn the prize based on the agreed upon coping plan.
  Arms: Child life standard of care + incentives provided with conditional agreement.
Behavioral: Child life standard of care + incentive provided unconditionally. — Patient is provided standard preparation and support provided to the participant by a Certified Child Life Specialist. After the procedure is complete the patient is provided with a prize. The patient does not need to do anything to earn the prize.
  Arms: Child life standard of care + incentive provided unconditionally.

SUMMARY:
The goal of this clinical trial is to learn about the use of incentives in pediatric patients requiring medical procedures. The main questions it aims to answer are: Are incentives effective at reducing pediatric anxiety for medical procedures? What is the best way to use incentives with pediatric populations requiring medical procedures? Participants will be provided support in preparation for their procedure and during the procedure by a child life specialist and might receive an incentive prize after their procedure. Participants distress levels during the procedure will be observed and they will be asked to rate their anxiety on a visual analog scale.

Researchers will compare the anxiety of those who did or did not receive an incentive after their procedure to see if incentives reduced procedural anxiety.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the impact incentives have on the distress and cooperation of children undergoing stressful medical procedures. The primary aim is to determine if offering an incentive reduces procedural distress for children undergoing stressful medical procedures. Secondly, if an incentive is offered does the process for offering the incentive (conditional or unconditional) to the patient impact the procedural distress of the patient. Patient anxiety and visit satisfaction will be looked at as secondary measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients and parent of patients aged 6-100 years who are undergoing a medical procedure
* Patients and parent of patients who are prepared and supported by a certified child life specialist.

Exclusion Criteria:

* Cognitive impairment that negates the use of the outcome tools
* Children younger than 6 years old, or older than 17 years old.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 187 (Estimated)
Dates: Start 2023-06-02 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
modified Yale Preoperative Anxiety Scale (mYPAS) | Immediately after the intervention/procedure/surgery
  Observational measure of anxiety in pediatric patients. Scores range from 23.33 to 100, lower scores meaning less anxiety.
Visual Scale Self-Report Anxiety | Immediately after the intervention/procedure/surgery
  Visual analog scale used for participants to report their perceived anxiety. Scores range from 0-100, lower scores meaning the participant is less anxious.

SECONDARY OUTCOMES:
Visit Satisfaction Survey | Immediately after the intervention/procedure/surgery
  Visit satisfaction survey completed by the accompanying parent.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Children's Hospital Colorado Anschutz, Aurora, Colorado
  - Children's Hospital Colorado North Campus, Broomfield, Colorado
  - Children's Hospital Colorado South Campus, Highlands Ranch, Colorado

IPD SHARING:
Plan to Share IPD: Undecided